CLINICAL TRIAL: NCT04740801
Title: Electrical Coupling Information From The RHYTHMIA HDx Mapping System and DIRECTSENSE Technology In The Treatment of Paroxysmal Atrial Fibrillation: A Non-Randomized Prospective Study With Contact Force
Brief Title: Electrical Coupling Information From The RHYTHMIA HDx Mapping System and DIRECTSENSE Technology In The Treatment of Paroxysmal Atrial Fibrillation (LOCALIZE CF)
Acronym: LOCALIZE CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM011
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PVI procedure (Other): Subjects will undergo ablation treatment of the pulmonary veins with the Rhythmia HDx mapping system with DirectSense technology. Subjects indicated for ablation treatment of de-novo PAF will be selected based on the inclusion/exclusion criteria and if deemed to be eligible for participation, will be asked to sign the Informed Consent Form. For all enrolled subjects who undergo the ablation procedure, the subjects will be treated with the commercial Rhythmia HDx System with commercially available Software Version 4.0.1 or greater (commercially approved version) with DIRECTSENSE™ and Force Computation Software Module; the IntellaMap Orion mapping catheter and the IntellaNav StablePoint ablation catheter.
  Interventions: Device: Ablation procedure

INTERVENTIONS:
Device: Ablation procedure — Catheter ablation of pulmonary veins with the Rhythmia HDx mapping system, IntellaMap Orion mapping catheter and IntellaNav StablePoint ablation catheter

SUMMARY:
The objective of this study is to evaluate whether local impedance (DIRECTSENSE™) drop on the INTELLANAV STABLEPOINT™ ablation catheter is associated with late pulmonary vein (PV) reconnections and durable conduction block in patients undergoing de novo PV isolation (PVI) for treatment of paroxysmal atrial fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

1. History of recurrent, symptomatic, paroxysmal atrial fibrillation (PAF), defined as atrial fibrillation (AF) that terminates spontaneously or with intervention (either procedure or drug therapy) within seven days of onset. Minimum documentation includes at least one AF episode electrocardiographically documented and at least one additional symptomatic recurrence with or without electrocardiographic documentation, within 365 days prior to enrollment.
2. Subjects who are eligible for an ablation procedure for paroxysmal AF according to international and local guidelines on catheter ablation of AF.
3. Subjects refractory or intolerant to at least one Beta Blocker, Calcium Channel Blocker, class I or III antiarrhythmic medication taken for the treatment of AF/AT (Atrial Tachycardia)/AFL (Atrial Flutter) or contraindicated to any class I or III antiarrhythmic medications, Beta Blocker or Calcium Channel Blocker.
4. Subjects who are willing and capable of providing informed consent.
5. Subjects who are willing and capable of participating in all testing associated with this clinical investigation at an approved clinical investigational center.
6. Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to local and national law.

Exclusion Criteria:

1. Any known contraindication to an AF ablation or anticoagulation
2. Continuous AF lasting longer than seven days from onset (no episodes within 365 days from enrollment)
3. History of previous LA ablation or surgical treatment for AF/AT/AFL
4. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
5. Subjects with life expectancy ≤ 6 months
6. Structural heart disease, heart conditions, or implanted devices as described below:

   1. Left ventricular ejection fraction < 35% based on the most recent imaging (≤ 180 days prior to enrollment)*
   2. LA diameter > 5.5 cm or LA volume >50 ml/m² indexed based on the most recent imaging (≤ 180 days prior to enrollment)*
   3. Heart failure with New York Heart Association (NYHA) Class III or IV
   4. Previous cardiac surgery (e.g. ventriculotomy or atriotomy, CABG, PTCA, stent procedure) within 90 days prior to enrollment
   5. Implantable cardiac device procedures (e.g. PM, ICD, CRT) within 30 days prior to enrollment
   6. Severe valvular disease or presence of a prosthetic - mechanical or biological - heart valve in the LA (not including valve repair and annular rings)
   7. Severe mitral valve regurgitation or stenosis
   8. Known or pre-existing severe pulmonary vein stenosis
   9. Interatrial baffle, closure device, patch, or patent foramen ovale (PFO) occluder
   10. Presence of LA appendage occlusion device
   11. Presence of any pulmonary vein stents
   12. Unstable angina or ongoing myocardial ischemia
   13. Previous myocardial infarction within 90 days prior to enrollment
   14. Vena cava embolic protection filter devices and/or known femoral thrombus;
   15. Known left atrial thrombus, myxoma, or intracardiac mural thrombus
7. History of blood clotting or bleeding disease
8. Any prior history of documented cerebral infarct, TIA, or systemic embolism [excluding a post-operative deep vein thrombosis (DVT)] ≤180 days prior to enrollment
9. Active systemic infection
10. Pregnant, lactating (current or anticipated during study follow up), or women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion)
11. Subjects who are currently enrolled in any other concurrent study, with the exception of local mandatory governmental registries and observational studies/registries, without written approval from the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Association between Local Impedance drop values and PV reconnections | 0-3 months
  Correlation between local impedance drop collected during the blinded index procedure and sites of late PV reconnection/durable block at 3-months.

SECONDARY OUTCOMES:
Association between Local Impedance drop values and acute PV reconnections | 0-1 month
  Correlation between local impedance drop collected during the blinded index procedure and sites of acute gaps/block after a 20-minute wait period.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Garcia Bolao, MD, Principal Investigator — Clinica Universitaria de Navarra; Hüseyin Ince, MD, Principal Investigator — Vivantes Klinikum am Urban; Francesco Solimene, MD, Principal Investigator — Casa Di Cura 'Montevergine' S.P.A.; Armin Luik, MD, Principal Investigator — Staedtisches Klinikum Karlsruhe
Locations (5):
- Germany (2):
  - Vivantes Klinikum Am Urban, Berlin
  - Städtisches Klinikum Karlsruhe, Karlsruhe
- Italy (2):
  - Casa di Cura Montevergine S.p.A., Mercogliano, Avellino
  - Centro Cardiologico Monzino, Milan
- Clinica Universidad de Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No
No requests for study data have been made at this time, however Boston's Scientific's policy on data sharing can be found at http:// www.bostonscientific.com/en-US/data-sharing-requests.html